CLINICAL TRIAL: NCT06345690
Title: VIA Disc NP Registry 3.0
Status: Recruiting | Type: Observational
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIA-2023-003
Record Dates: First submitted 2024-03-06; First posted 2024-04-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Discogenic Pain; Back Pain; Back Pain, Low
Keywords: Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VIA Disc NP: Patients meeting study criteria receiving Vivex VIA Disc NP injection as treatment
  Interventions: Other: VIA Disc NP

INTERVENTIONS:
Other: VIA Disc NP — VIA Disc NP - Allograft tissue injection

SUMMARY:
Registry is to observe and trend patterns of care and outcomes for patients treated with VIA Disc NP.

DETAILED DESCRIPTION:
The Registry is intended to collect data for patients having received treatment with VIA Disc NP.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol
2. 18 years of age or older
3. Literate, able to speak and read English, and able to complete questionnaires independently
4. Subject received a VIA Disc NP injection with 1 or more levels within 90 days of the baseline visit.

Exclusion Criteria:

1. Participant did not receive VIA Disc NP injection
2. Participant is pregnant (self-reported, no special study pregnancy testing needed).
3. Any contraindications as noted in the VIA Disc NP Instructions for Use
4. Previous treatment with VIA Disc NP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with and treated for back pain.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 1, 3, 6, & 12 months
  Change in Numeric Rating Scale (NRS) scores. Eleven point pain scale used for patient self-reporting of back pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable).
Oswestry Disability Index (ODI) | 1, 3, 6, & 12 months
  Change in scores from Oswestry Disability Index (ODI). An index comprising of ten categories of function to quantify disability due to back pain.
Patient Satisfaction | 1, 3, 6, & 12 months
  Patient reported assessment of treatment regarding their experience with the procedure. Four different responses, which range from Not at all satisfied (worst) to Extremely Satisfied (best).
Frequency of Pain Medication Use | 1, 3, 6, & 12 months
  Assesses the frequency and type of pain medication administered to participants at baseline and follow-up visits scheduled at 1, 3, 6, and 12 months. Data will be collected to track changes in pain medication usage over time.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Zaccari, Study Director — Sponsor - Vivex Biologics
Locations (26):
- United States (26):
  - Mocek Spine, Little Rock, Arkansas
  - MD Pain, Englewood, Colorado
  - Western Rockies Interventional Pain, Grand Junction, Colorado
  - The Denver Spine & Pain Institute, Greenwood Village, Colorado
  - Premier Spine and Pain Institute, Thornton, Colorado
  - The Orthopedic Institute, Gainesville, Florida
  - Raso Pain Center, Jupiter, Florida
  - Interventional Spine Care of the Palm Beaches, West Palm Beach, Florida
  - Horizon Clinical Research, Jasper, Georgia
  - The Orthopedic Research Foundation, Inc., Fishers, Indiana
  - Interventional Pain Specialists - Pain Clinic, Opelousas, Louisiana
  - Paradigm Health System, Slidell, Louisiana
  - Premier Pain Solutions, Asheville, North Carolina
  - Comprehensive Pain Consultants of the Carolinas, Hendersonville, North Carolina
  - Crystal Coast Pain Management, Morehead City, North Carolina
  - Crystal Coast Pain Management, New Bern, North Carolina
  - Align Interventional Pain, Edmond, Oklahoma
  - Fox Chase Pain Management_Delaware Valley Pain and Spine Institute (DVPSI), Trevose, Pennsylvania
  - Atlantic Coast Spine & Pain, Conway, South Carolina
  - Renew Pain Solutions, Greenville, South Carolina
  - Specialists in Pain Managment, Chattanooga, Tennessee
  - Freedom Spine, Boerne, Texas
  - Corpus Chrisi Pain Medicine, Corpus Christi, Texas
  - Advanced Spine and Pain Center, San Antonio, Texas
  - Pain and Wellness Institute of Texas, Spring Branch, Texas
  - Precision Spine Care, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No